CLINICAL TRIAL: NCT07275580
Title: Effectiveness of Short-Course Antibiotic Prophylaxis After Simple Tooth Extraction in Immunosuppressed Patients With Autoimmune Rheumatic Diseases
Brief Title: Antibiotic Prophylaxis After Simple Tooth Extraction in Immunosuppressed Patients With Autoimmune Rheumatic Diseases
Acronym: PRO-EXOD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 69108723.1.0000.0068
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Rheumatic Diseases; Tooth Extraction; Infection Prevention; Antibiotic Prophylaxis
Keywords: Autoimmune Rheumatic Diseases; Tooth Extraction; Infection Prevention; Amoxicillin; Antibiotic Stewardship
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Antibiotic Prophylaxis (Active Comparator): Single 2 g oral dose administered 30-60 minutes before tooth extraction
  Interventions: Drug: Amoxicillin
- Arm 2 - No Antibiotic Prophylaxis (Placebo Comparator): Four matching placebo tablets administered 30-60 minutes before extraction
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin 2 g a single prophylactic dose prior to simple extraction.
  Arms: Arm 1 - Antibiotic Prophylaxis
Other: Placebo — Matching placebo tablets administered as a single dose prior to extraction
  Arms: Arm 2 - No Antibiotic Prophylaxis

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate whether single-dose amoxicillin prophylaxis administered prior to simple tooth extraction reduces postoperative infection rates in immunosuppressed patients with autoimmune rheumatic diseases (ARDs).

Although antibiotic prophylaxis is not recommended for healthy individuals undergoing simple extractions, immunosuppressed ARD patients frequently receive antibiotics despite limited evidence supporting this practice.

Secondary objectives include assessing infection severity, postoperative complications, and the impact of ARD diagnosis and immunosuppressive treatment on infection risk.

DETAILED DESCRIPTION:
Simple tooth extractions are common procedures, and postoperative infection rates are low in the general population. Current guidelines discourage prophylactic antibiotic use to reduce microbial resistance, adverse reactions, and microbiome disruption.

However, immunosuppressed patients with ARDs often receive prophylaxis due to theoretical risks of delayed healing and increased susceptibility to infection. Evidence in other immuno-compromised populations suggests that simple extractions may be safe without antibiotics, but no prospective trials have evaluated this issue specifically in ARD patients.

This study is the first prospective, randomized, double-blind, placebo-controlled trial designed to determine whether antibiotic prophylaxis is necessary in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of an ARD: SLE, RA, JIA, AS, PsA, IIM, systemic vasculitis, primary Sjögren's syndrome, or SSc
* Under immunosuppressive or biologic therapy ≥3 months
* Indication for simple extraction of tooth with chronic odontogenic focus
* Provided informed consent

Exclusion Criteria:

* Individuals who do not agree to participate in the study will be excluded.
* Patients who require more technically complex extractions, such as impacted or impacted third molars.
* Patients with local and systemic changes that require more extensive antibiotic coverage, such as cases with clinical signs of acute infections, anticoagulated patients, heart patients, patients who have undergone radiotherapy or are undergoing treatment for neoplasms.
* Patients allergic to amoxicillin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2029-01-17 (Estimated); Study Completion 2029-02-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of postoperative infections | 7 days post-extraction
  Proportion of participants developing postoperative infection, defined as purulent/serous exudate, fever (>37.8°C), or clinical signs of local infection.

SECONDARY OUTCOMES:
Severity and Duration of Infection | 7 days
  Presence and duration of purulent/serous exudate, fever (>37.8°C), or clinical signs of local infection and systemic symptoms
Incidence of Postoperative Complications | 7 days
  Presence of alveolitis, fever, edema, erythema, trismus, exudate, and pain
Influence of ARD Diagnosis and Immunosuppressive Regimen | 7 days
  Infection rate and severity related to ARD Diagnosis and Immunosuppressive Regimen
Disease Activity Flares | Day 1 through Day 30
  Disease Activity Flares according to specific ARD definitions of exacerbation, as follows:
  Systemic Lupus Erythematosus(SLE): Increase >3 points in SLE Disease Activity Index 2000(SLEDAI-2K) Rheumatoid Arthritis(RA): Increase in Disease Activity Score-C-reactive protein(DAS28-CRP)>1.2, or >0.6 if baseline DAS28-CRP>3.2 Juvenile Idiopathic Arthritis(JIA): Increase in JIA Disease Activity Score(JADAS-27) >5 points, or worsening ≥2 active joints Ankylosing Spondylitis(AS): Increase in AS Disease Activity Score(ASDAS) >0.9. Psoriatic Arthritis(PsA): Worsening in Disease Activity Index for PsA(DAPSA) Systemic Vasculitis: Increase in Birmingham Vasculitis Activity Score(BVAS). Primary Sjögren's Syndrome: EULAR Sjögren's Syndrome Disease Activity Index(ESSDAI) Systemic Sclerosis (SSc): Increase in modified Rodnan skin score, new digital ulcers, worsening dyspnea, or increase in EULAR Systemic Sclerosis Impact of Disease Index (ScleroID) Inflammatory Myopathies (IIM): muscle weakness, CK

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa Bonfá, Full Professor, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da USP - HCFMUSP

IPD SHARING:
Plan to Share IPD: No